CLINICAL TRIAL: NCT03826771
Title: Post-Stroke Optimization of Walking Using Explosive Resistance: Concurrent Effects on Depression (POWER-D Trial)
Brief Title: Post-Stroke Optimization of Walking Using Explosive Resistance
Acronym: POWER-D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00077223; R01HD095137 (NIH)
Record Dates: First submitted 2019-01-29; First posted 2019-02-01 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Depression
Keywords: stroke; rehabilitation; depression; exercise
MeSH Terms: conditions — Stroke; Depression; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POWER training (Experimental): high velocity strength training
  Interventions: Behavioral: Power training
- Stretching (Active Comparator): Upper and lower body range of motion exercises
  Interventions: Behavioral: Stretching

INTERVENTIONS:
Behavioral: Power training — high-intensity lower extremity resistance training
  Arms: POWER training
Behavioral: Stretching — upper and lower body range of motion exercises
  Arms: Stretching

SUMMARY:
The investigators will study the effects of a 12 week strength training program on individuals who have had a stroke and are depressed to see if this type of exercise training helps treat depression and improves walking function. Our goal is to use the information collected in this study to help design treatments for people who have had a stroke that will help with many of the common consequences of stroke, including depression, muscle weakness and slow walking. Progress toward overcoming some of these issues would be incredibly valuable to any person who has had a stroke and their families.

DETAILED DESCRIPTION:
Depression is the most common neuropsychiatric manifestation following stroke and current treatments are largely ineffective. Depression has both direct and indirect effects on response to rehabilitation, thus subjects with post-stroke depression (PSD) are routinely excluded from clinical trials and treatment options are extremely limited. The investigators propose to determine the impact of a novel, high-intensity resistance training program, Post-stroke Optimization of Walking using Explosive Resistance (POWER) training, on post-stroke depressive symptoms. Further, the investiators will determine if depression limits training-induced improvements in muscular and locomotor function. This project is based on the premise that depression negatively affects the potential for neuroplastic changes to occur in response to treatment such that rehabilitation may not produce the same adaptations that it does in non-depressed individuals. The investigators propose that effective treatment for PSD would result in a virtuous cycle where reducing depression enhances neuroplastic changes, thereby facilitating functional gains. That is, effectively treating depression will make the individual better able to recover from stroke. Furthermore, in addition to its beneficial effects on depression, POWER training is known to improve post-stroke walking, thus providing an attractive option for treating depression as well as an established vehicle to study the effects of PSD on response to rehabilitation. The experiments proposed as part of this project are designed to address critical questions related to 1) the effects of POWER training on depressive symptoms; 2) the potential for PSD to limit improvements following training; and 3) the interaction between improvements in depression and increases in walking function. Successful completion of this project will provide a foundation for larger scale trials to determine dosing parameters as well as establish therapeutic effectiveness of POWER training on post-stroke depression as well as identify the mechanisms that may be responsible for the changes that occur in response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* age 50-70
* stroke within the past 6 to 60 months
* residual paresis in the lower extremity (Fugl-Meyer LE motor score <34)
* ability to walk without assistance and without an AFO during testing and training at speeds ranging from 0.2-0.8 m/s
* no antidepressant medications or no change in doses of psychotropic medication for at least 4 weeks prior to the study (6 weeks if newly initiated medication)
* HRSD question #9 regarding suicide <2; and 7) provision of informed consent.

Exclusion Criteria:

* Unable to ambulate at least 150 feet prior to stroke, or experienced intermittent claudication while walking
* history of congestive heart failure, unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during ADL's
* History of COPD or oxygen dependence
* Preexisting neurological disorders, dementia or previous stroke
* History of major head trauma
* Legal blindness or severe visual impairment
* history of psychosis or other Axis I disorder that is primary
* Life expectancy <1 yr.
* Severe arthritis or other problems that limit passive ROM
* History of DVT or pulmonary embolism within 6 months
* Uncontrolled diabetes with recent weight loss, diabetic coma, or frequent insulin reactions
* Severe hypertension with systolic >200 mmHg and diastolic >110 mmHg at rest
* attempt of suicide in the last 2 years or at suicidal risk assessed by SCID interview
* History of seizures or currently prescribed anti-seizure medications
* Current enrollment in a clinical trial to enhance motor recovery
* Pregnancy

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- POWER Training - Depressed: high velocity strength training for depressed individuals
  Power training: high-intensity lower extremity resistance training
- POWER Training - Non-Depressed: high velocity strength training for non-depressed individuals
  Power training: high-intensity lower extremity resistance training
Period: Overall Study
Arm/Group | POWER Training - Depressed | Stretching | POWER Training - Non-Depressed
Started | 19 | 12 | 17
Completed | 12 | 9 | 15
Not Completed | 7 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- POWER Training - Depressed: high velocity strength training in depressed individuals
  Power training: high-intensity lower extremity resistance training
- POWER Training - Non-Depressed: high velocity strength training in non-depressed individuals
  Power training: high-intensity lower extremity resistance training
- Total: Total of all reporting groups
Arm/Group | POWER Training - Depressed | Stretching | POWER Training - Non-Depressed | Total
Number analyzed (Participants) | 19 | 12 | 17 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 8 | 8 | 32
  >=65 years | 3 | 4 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.37 (10.82) | 57.83 (12.25) | 62.59 (9.8) | 56.96 (11.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 4 | 22
  Male | 9 | 4 | 13 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 7 | 5 | 18
  White | 12 | 5 | 12 | 29
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Score of Depression as Assessed by the Hamilton Rating Scale for Depression
Description: The HAM-D is a clinician-rated scale with scores based on clinical interview and family report. It addresses both somatic and psychological symptoms of depression. Items are rated on either a 5-point scale (0 to 4) or 3-point scale (0 to 2), where higher scores represent increasing severity of depression. The scores of the 17 items are summed to obtain a total score (minimum score: 0, maximum score: 52).
Time Frame: Visit 1 through visit 24 (up to 12 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | POWER Training - Depressed | Stretching | POWER Training - Non-Depressed
Number analyzed (Participants) | 14 | 9 | 15
units on a scale | 5.20 (4.31) | 2.17 (4.72) | 0.14 (2.83)

2. Secondary Outcome: Change in Self Selected Walking Speed
Description: Subjects will walk on a 14-ft. long gait mat (GaitRite) to measure self-selected and fastest comfortable walking speed and other spatiotemporal parameters of walking. Subjects will be permitted a practice trial, and then be asked to complete three trials at each speed. For all trials, subjects will wear their own shoes and be asked to walk without an assistive device or ankle-foot orthosis.
Time Frame: Visit 1 through visit 24 (up to 12 weeks)
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | POWER Training - Depressed | Stretching | POWER Training - Non-Depressed
Number analyzed (Participants) | 14 | 9 | 15
meters per second | 0.08 (0.02) | 0.06 (0.02) | 0.21 (0.06)

ADVERSE EVENTS:
Time Frame: throughout the 12 week training intervention
Arm/Group | POWER Training - Depressed | Stretching | POWER Training - Non-Depressed
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/12 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/12 | 0/17
Other Adverse Events (participants affected / at risk) | 2/19 | 0/12 | 1/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | POWER Training - Depressed (N=19) | Stretching (N=12) | POWER Training - Non-Depressed (N=17)
mild injury (sprain/contusion) (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-23): https://cdn.clinicaltrials.gov/large-docs/71/NCT03826771/Prot_SAP_000.pdf